CLINICAL TRIAL: NCT05633368
Title: Impact of Covid-19 Pandemic on Patients With Unipolar Depressive Disorder: Effects of Discontinuing Continuation or Maintenance Electroconvulsive Therapy
Brief Title: Impact of Covid-19 Pandemic on Patients Receiving Continuation or Maintenance Electroconvulsive Therapy
Acronym: COVID-M-ECT
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: BC-07543
Record Dates: First submitted 2020-06-29; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Electroconvulsive Therapy; Major Depressive Disorder; Covid-19
Keywords: Electroconvulsive therapy; Maintenance ECT; Continuation ECT; Major depressive disorder; Covid-19
MeSH Terms: conditions — Depressive Disorder, Major; COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Discontinuation of C/M-ECT: Participants with major depressive disorder who are unable to continue maintenance (M-ECT) or continuation electroconvulsive therapy (C-ECT) due to hospital restrictions during Covid-19 or due to personal preference.
  Interventions: Other: Questionnaires
- Continuation of C/M-ECT: Participants with major depressive disorder who are able to continue maintenance (M-ECT) or continuation electroconvulsive therapy (C-ECT) during Covid-19.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will be contacted every three weeks to assess depressive symptomatology and possible relapse.
  * Patient Health Questionnaire (PHQ-9)
  * Clinical Global Impression (CGI)
  * Scaling question regarding depressive symptomatology

SUMMARY:
Electroconvulsive therapy is a safe and effective therapeutic strategy in patients with treatment resistant depression. As relapse after successful ECT is significant even with adequate pharmacological strategies, continuation (up to 6 months after completion of index-ECT) or maintenance ECT (more than 6 months after index-ECT) is often necessary to maintain remission. During the current Covid-19 pandemic hospitals redirected resources and closed or significantly diminished ECT services. In this study we aim to assess the impact of discontinuing maintenance electroconvulsive therapy in patients diagnosed with unipolar depressive disorder.

DETAILED DESCRIPTION:
During the height of the Covid-19 pandemic in Belgium all patients receiving continuation or maintenance electroconvulsive therapy (ECT) for major depressive disorder in two ECT centers in Belgium will be included. Due to differences in Covid-19 infection rates and hospital management decisions, one ECT-service temporarily halted all electroconvulsive treatments, where as the other ECT-service continued continuation and maintenance treatments. Depressive symptomatology and relapse rates will be assessed during the diminished accessibility of electroconvulsive treatment.

ELIGIBILITY:
Inclusion Criteria:

* Continuation or maintenance ECT, in treatment at two specified ECT-centers in Belgium
* Unipolar depressive disorder

Exclusion Criteria:

* Unable to provide informed consent
* Unable to comply with study requirements (telephone questionnaire)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving continuation or maintenance ECT for unipolar depressieve disorder in two ECT clinics in Belgium at the time of the start of the study (31/03/2020).
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Change in depressive symptoms (PHQ-9) | From time of inclusion until maximum 9 months (or sooner if resumption of ECT)
  Change in depressive symptoms as measured by the patient health questionnaire via phone or through direct participant contact. The PHQ is a 9-question instrument to screen for the presence and severity of depression. The minimum score is 0 and the maximum score is 27, with a higher score indicating more depressive symptoms.
Change in depressive symptoms, subjective score, scaling question | From time of inclusion until maximum 9 months (or sooner if resumption of ECT)
  Change in depressive symptoms as measured by the following scaling question: How would you rate your depressive symptoms on a scale from 0 to 10 with 0 indicating no depressive symptoms and 10 indicating extremely severe depressive symptoms'.
Change in depressive symptoms, subjective score | From time of inclusion until maximum 9 months (or sooner if resumption of ECT)
  Change in depressive symptoms as measured by the patient-rated question: 'How would you describe the severity of your depressive symptoms?'. No depressive symptoms equals a score of 0 and severe depressive symptoms equals a score of 3.
Change in depressive symptoms (CGI) | From time of inclusion until maximum 9 months (or sooner if resumption of ECT)
  Change in depressive symptoms as measured by the Clinical Global impression Scale. This is a clinician-rated scale to assess severity and change in symptomatology with a score of 1 indicating normal or no illness or very much improved and 7 severly ill or very much deteriorated.
Relapse, depression | From time of inclusion until maximum 9 months (or sooner if resumption of ECT)
  During every study contact the need for restart of electroconvulsive treatment or hospital admission will be evaluated by the investigator. If ECT restart or hospital admission is advised, this will be an indication of relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Nele Van de Velde, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent, East-Flanders
  - AZ Groeninge, Kortrijk, West-Flanders

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are not publicly available due to confidentiality issues but are available from the corresponding author upon reasonable request.